CLINICAL TRIAL: NCT05657145
Title: Visualization of the Papilla Through Use of the NuView Device in Patients With FAP
Acronym: NuView
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Keith Obstein, Professor, Vanderbilt University Medical Center
Other Study IDs: NuView_220899
Record Dates: First submitted 2022-12-01; First posted 2022-12-20 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Familial Adenomatous Polyposis
MeSH Terms: conditions — Adenomatous Polyposis Coli

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Familiar Adenomatous Polyposis: All patient in this group will have the NuView device used to assist in the visualization of the papilla.

SUMMARY:
The goal of this observational study is to test the NuView device in participants with familial adenomatous polyposis (FAP). The main question it aims to answer is:

* can the papilla be visualized using a forward-facing endoscope outfitted with the NuView device. Participants will undergo standard of care esophagogastroduodenoscopy with an additional endoscopic exam using NuView device, for which participant have given prior consent.

DETAILED DESCRIPTION:
The clinical practice at Vanderbilt University Medical Center will first perform the routine upper endoscopic exam with a forward-viewing gastroscope to evaluate the patient's esophagus, stomach, and duodenum. After this has been completed, the forward-viewing endoscope will be removed from the patient and outfitted with the EndoTheia NuView. The endoscope with NuView will then be inserted transorally down the esophagus, traverse the stomach, and be passed into the duodenum for visualization of the papilla. After the papilla is visualized, the endoscope with NuView will be removed from the patient. As per standard of care, the conventional side-viewing endoscope will then be inserted transorally down the esophagus, traverse the stomach, and be passed into the duodenum for visualization of the papilla. The side-viewing endoscope will then be removed from the patient. The Investigators plan to enroll 3 FAP patients who are already scheduled to undergo their standard of care endoscopic exam. The primary endpoint of the study is successful visualization of the papilla with the NuView platform.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 to 70 years of age.
* Able to provide written informed consent.
* Have FAP

Exclusion Criteria:

* Females who are pregnant. As part of routine pre-operative care, all females of childbearing potential will undergo either urine or blood pregnancy testing.
* Cancer positive subjects or any patients currently undergoing any treatment or therapy to treat, cure, or mitigate cancer.
* Patients who do not meet inclusion criteria
* Patients who are unable or unwilling to provide informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential subjects will be identified from patients in the Vanderbilt University Medical Center Digestive Disease Center who are scheduled to undergo their endoscopic screening for FAP. FAP is a hereditary condition in which a person develops numerous precancerous polyps, called adenomas, within the small and large intestine. Currently, it is recommended that FAP patients undergo serial endoscopic exams to assess the colon for polyp formation every year and every 2-3 years to look for adenomas in the small intestine-specifically on the duodenal papilla.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2023-01-27 (Actual); Primary Completion 2025-12-30 (Actual); Study Completion 2025-12-30 (Actual)

PRIMARY OUTCOMES:
Visualization of papilla | 1 day
  Successful visualization of the papilla with a standard gastroscope equipped with the NuView platform.

CONTACTS AND LOCATIONS:
Overall Officials: Keith L Obstein, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2022-05-05): https://cdn.clinicaltrials.gov/large-docs/45/NCT05657145/Prot_000.pdf
  • Informed Consent Form (2022-08-02): https://cdn.clinicaltrials.gov/large-docs/45/NCT05657145/ICF_001.pdf